CLINICAL TRIAL: NCT01582061
Title: An Open-label, Multi-center, Expanded Access Study of Pasireotide s.c. in Patients With Cushing's Disease (Seascape).
Brief Title: An Open-label, Multi-center, Expanded Access Study of Pasireotide s.c. in Patients With Cushing's Disease.
Acronym: SEASCAPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230B2406
Record Dates: First submitted 2012-04-12; First posted 2012-04-20 (Estimated); Results first posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Cushing's Disease
Keywords: Cushing's disease; Hormone disorder; Cortisol; Adrenocorticotropic hormone; Pituitary tumor; SOM230; adult
MeSH Terms: conditions — Pituitary ACTH Hypersecretion; Pituitary Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pasireotide 600 μg (Experimental): Pasireotide sub-cutaneous was supplied in 1 ml ampoules containing 600 μg pasireotide per 1 ml of solution and was administered BID. Starting dose was 600 μg for glucose impaired metabolism patients. Mean daily dose category is defined on the mean daily dose considering the following grouping rule: 600 μg bid group includes all patients whose mean daily dose < 1500 μg /day.
  Interventions: Drug: Pasireotide sub-cutaneous
- Pasireotide 900 μg (Experimental): Pasireotide sub-cutaneous was supplied in 1 ml ampoules containing 900 μg pasireotide per 1 ml of solution and was administered BID. Starting dose was 900 μg. Mean daily dose category is defined on the mean daily dose considering the following grouping rule: 900 μg bid group includes all patients whose mean daily dose ≥ 1500 μg /day
  Interventions: Drug: Pasireotide sub-cutaneous

INTERVENTIONS:
Drug: Pasireotide sub-cutaneous — Pasireotide sub-cutaneous was supplied in 1 ml ampoules containing 900 μg, 600 μg, or 300 μg pasireotide per 1 ml of solution and was administered BID. Starting dose was 900 μg and 600 μg for glucose impaired metabolism patients
  Other Names: SOM230 sub-cutaneous

SUMMARY:
This study provided access to pasireotide sc in patients with Cushing's disease.and provided additional information for safety and efficacy of pasireotide s.c.

DETAILED DESCRIPTION:
Purpose of this study was to give access to pasireotide sc for patients with Cushing's disease as no medical treatment for Cushing's disease was approved at the time of the study initiation. The study population consisted of patients with persistent or recurrent Cushing's disease or patients with de novo Cushing's disease that were not considered candidates for pituitary surgery (poor surgery candidates, surgically unapproachable tumor, patients with no visible pituitary tumor, patients who refused surgery). A confirmed Cushing's disease diagnosis was required.

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent obtained prior to any screening procedures
2. Male or female patients aged 18 years or greater
3. Patients with confirmed diagnosis of Cushing's disease as evidenced by mean urinary free cortisol of three 24-hour urine samples collected during the 3-week screening period above the upper limit of the laboratory normal range morning plasma ACTH within the normal or above normal range either MRI confirmation of pituitary adenoma (greater than or equal to 0.6 cm), or inferior petrosal sinus gradient >3 after CRH stimulation for those patients with a microadenoma less than 0.6 cm, or for patients who have had prior pituitary surgery, histopathology confirming an ACTH staining adenoma.
4. Patients with de novo Cushing's disease must not be considered as candidates for pituitary surgery (i.e. poor surgical candidates, surgically unapproachable tumors, patients with no visible pituitary tumor, patients who refuse to have surgical treatment)
5. Karnofsky performance status >60 (i.e. requires occasional assistance, but is able to care for most of his personal needs)
6. For patients on previous medical treatment for Cushing's disease the following washout periods must be completed before screening assessments are performed

   * Inhibitors of steroidogenesis (e.g. ketoconazole, metyrapone, rosiglitazone): 1 week
   * Dopamine agonists (e.g. bromocriptine, cabergoline): 4 weeks
   * Mitotane: 6 months
   * Octreotide LAR and Lanreotide autogel: 8 weeks
   * Lanreotide SR: 4 weeks
   * Octreotide (immediate release formulation): 1 week
   * Glucocorticoid receptor inhibitor (mifepristone): 4 weeks

Exclusion criteria:

1. Radiotherapy of the pituitary <4 weeks before screening or patient who has not recovered from side effects
2. Patients with compression of the optic chiasm causing acute clinically significant visual field defect
3. Patients with Cushing's syndrome due to ectopic ACTH secretion
4. Patients with hypercortisolism secondary to adrenal tumors or nodular (primary) bilateral adrenal hyperplasia
5. Patients who have a known inherited syndrome as the cause for hormone over secretion (i.e. Carney Complex, McCune-Albright syndrome, MEN-1)
6. Patients with a diagnosis of glucocorticoid-remedial aldosteronism (GRA)
7. Patients who have undergone major surgery within 1 month prior to screening
8. Patients with known gallbladder or bile duct disease, acute or chronic pancreatitis (patients with asymptomatic cholelithiasis and asymptomatic bile duct dilation can be included)
9. Diabetic patients whose blood glucose is poorly controlled as evidenced by HbA1C >8%
10. Patients who have clinically significant impairment in cardiovascular function or are at risk thereof, as evidenced by congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, clinically significant bradycardia, high grade AV block, history of acute MI less than one year prior to study entry

    * QTcF >450 msec at screening
    * History of syncope or family history of idiopathic sudden death
    * Risk factors for Torsades de Pointes such as uncorrected hypokalemia, uncorrected hypomagnesemia, cardiac failure
    * Concomitant disease(s) that could prolong the QT interval such as autonomic neuropathy (caused by diabetes or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism, concomitant medication(s) with known risk for TdP
11. Patients with liver disease or history of liver disease such as cirrhosis, chronic active hepatitis B and C, or chronic persistent hepatitis, or patients with ALT or AST more than 2 x ULN, serum creatinine >2.0 x ULN, serum bilirubin >1.5 x ULN, serum albumin < 0.67 x LLN at screening
12. Patients who have any current or prior medical condition that can interfere with the conduct of the study or the evaluation of its results, such as

    * History of immunocompromise, including a positive HIV test result (Elisa and Western blot). An HIV test will not be required, however, previous medical history will be reviewed
    * Presence of active or suspected acute or chronic uncontrolled infection
    * History of, or current alcohol misuse/abuse in the 12 month period prior to screening
13. Female patients who are pregnant or lactating, or are of childbearing potential and not practicing a medically acceptable method of birth control. If a woman is participating in the trial then one form of contraception is sufficient (pill or diaphragm) and the partner should use a condom. If oral contraception is used in addition to condoms, the patient must have been practicing this method for at least two months prior to screening and must agree to continue the oral contraceptive throughout the course of the study and for one month after the study has ended. Male patients who are sexually active are required to use condoms during the study and for three month afterwards as a precautionary measure (available data do not suggest any increased reproductive risk with the study drugs)
14. Patients who have participated in any clinical investigation with an investigational drug within 1 month prior to screening or patients who have previously been treated with pasireotide
15. Known hypersensitivity to somatostatin analogues
16. Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will be unable to complete the entire study
17. Patients with presence of Hepatitis B surface antigen (HbsAg)
18. Patients with presence of Hepatitis C antibody test (anti-HCV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-08-16 (Actual); Primary Completion 2017-01-26 (Actual); Study Completion 2017-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (58):
- United States (17):
  - Advanced Research, LLC, Peoria, Arizona
  - St Josephs Hospital & Medical Center St Joes, Phoenix, Arizona
  - University of California at Los Angeles UCLA Tiverton, Los Angeles, California
  - LA Biomedical Research at Harbor UCLA Medical Center, Torrance, California
  - Emory University School of Medicine, Atlanta, Georgia
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - Diabetes and Endocrinology Associates, PC, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of New Mexico Hospital UNM, Albuquerque, New Mexico
  - Mount Sinai School of Medicine, New York, New York
  - Oregon Health and Science University OHSU 5, Portland, Oregon
  - University of Pennsylvania Medical Center Univ Penn, Philadelphia, Pennsylvania
  - Allegheny Endocrinology Associates, Pittsburgh, Pennsylvania
  - Mid South Endocrine Associates, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Swedish Cancer Institute Swedish Cancer Institute (SC), Seattle, Washington
- Brazil (6):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Londrina, Paraná
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Joinville, Santa Catarina
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Prague, Czech Republic, Czechia
- Germany (14):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Würzburg
- Greece (4):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Novartis Investigative Site, El Achrafiyé, Lebanon
- Romania (3):
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Iași
- Novartis Investigative Site, Moscow, Russia
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (7):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Ourense, Galicia
  - Novartis Investigative Site, Pontevedra, Galicia
  - Novartis Investigative Site, Valencia, Valencia
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Songkhla

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fleseriu M, Iweha C, Salgado L, Mazzuco TL, Campigotto F, Maamari R, Limumpornpetch P. Safety and Efficacy of Subcutaneous Pasireotide in Patients With Cushing's Disease: Results From an Open-Label, Multicenter, Single-Arm, Multinational, Expanded-Access Study. Front Endocrinol (Lausanne). 2019 Jul 16;10:436. doi: 10.3389/fendo.2019.00436. eCollection 2019. PMID 31379734

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After a 21-day screening period, patients who met the inclusion/exclusion criteria received pasireotide subcutaneous twice a day (BID)
Period: Overall Study
Arm/Group | Pasireotide 600 μg | Pasireotide 900 μg
Started | 49 | 55
Completed | 21 | 19
Not Completed | 28 | 36
Not completed — Lack of Efficacy | 3 | 23
Not completed — Adverse Event | 12 | 8
Not completed — Withdrawal by Subject | 10 | 4
Not completed — Abnormal laboratory value(s) | 1 | 0
Not completed — Death | 0 | 1
Not completed — condition no longer requires study drug | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pasireotide 600 μg | Pasireotide 900 μg | Total
Number analyzed (Participants) | 49 | 55 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (13.14) | 39.9 (12.55) | 42.5 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 47 | 84
  Male | 12 | 8 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 15 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 39 | 36 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a Drug-related Adverse Event That is Recorded as Grade 3 or 4 or as a Serious Adverse Event (SAE)
Description: Only AEs occurring on or after the start of study treatment and no more than 28 days after the discontinuation of study treatment. A patient with multiple occurrences of an AE under one treatment is counted only once in the AE category for that treatment. A patient with multiple severity grades for an AE while on a treatment, is only counted under the maximum grade.
Time Frame: Baseline up to approximately 256 weeks
Population: Three additional arms were created to display subset of subjects with specific criteria.
Measure: Number; unit: percentage of participants
Groups:
- 600 µg Bid - All Grades: All grades of adverse events. Pasireotide sub-cutaneous was supplied in 1 ml ampoules containing 600 μg pasireotide per 1 ml of solution and was administered BID. Starting dose was 600 μg for glucose impaired metabolism patients. Mean daily dose category is defined: 600 μg bid group includes all patients whose mean daily dose < 1500 μg /day.
- 600 μg - Grades 3/4: Adverse event grades 3 and 4. Pasireotide sub-cutaneous was supplied in 1 ml ampoules containing 600 μg pasireotide per 1 ml of solution and was administered BID. Starting dose was 600 μg for glucose impaired metabolism patients
- 900 μg - All Grades: All grades of adverse events. Pasireotide sub-cutaneous was supplied in 1 ml ampoules containing 900 μg pasireotide per 1 ml of solution and was administered BID. Starting dose was 900 μg. Mean daily dose category is defined : 900 μg bid group includes all patients whose mean daily dose ≥ 1500 μg /day
- 900 μg - Grades 3/4: Adverse event grades 3 and 4. Pasireotide sub-cutaneous was supplied in 1 ml ampoules containing 900 μg pasireotide per 1 ml of solution and was administered BID. Starting dose was 900 μg
- All Patients - All Grades; All Patients - Grades 3/4: All grades of adverse events for all patients who received 600 µg bid or 900 µg bid of pasireotide sub-cutaneous.
Arm/Group | 600 µg Bid - All Grades | 600 μg - Grades 3/4 | 900 μg - All Grades | 900 μg - Grades 3/4 | All Patients - All Grades | All Patients - Grades 3/4
Number analyzed (Participants) | 49 | 49 | 55 | 55 | 104 | 104
percentage of participants
  Any primary system organ class | 53.1 | 53.1 | 29.1 | 27.3 | 40.4 | 39.4
  Metabolism and nutrition disorders: number analyzed (Participants) | 49 | 26 | 55 | 55 | 104 | 104
  Metabolism and nutrition disorders | 26.5 | 26.5 | 12.7 | 10.9 | 19.2 | 18.3
  Gastrointestinal disorders | 18.4 | 18.4 | 7.3 | 7.3 | 12.5 | 12.5
  Investigations | 8.2 | 8.2 | 3.6 | 3.6 | 5.8 | 5.8
  Hepatobiliary disorders | 2.0 | 2.0 | 5.5 | 5.5 | 3.8 | 3.8
  Endocrine disorders | 6.1 | 6.1 | 0 | 0 | 2.9 | 2.9
  Gen disorders,admin site conditions | 4.1 | 4.1 | 0 | 0 | 1.9 | 1.9
  Ear and labyrinth disorders | 2.0 | 2.0 | 0 | 0 | 1.0 | 1.0
  Infections and infestations | 2.0 | 2.0 | 0 | 0 | 1.0 | 1.0
  Musculoskeletal and connective tissue disorders | 2.0 | 2.0 | 0 | 0 | 1.0 | 1.0
  Neoplasms benign, malignant and unspecified | 2.0 | 2.0 | 0 | 0 | 1.0 | 1.0
  Nervous system disorders | 2.0 | 2.0 | 0 | 0 | 1.0 | 1.0
  Psychiatric disorders | 0 | 0 | 1.8 | 1.8 | 1.0 | 1.0
  Respiratory, thoracic, mediastinal disorders | 0 | 0 | 1.8 | 0 | 1.0 | 0

2. Secondary Outcome: Percentage of Patients With Mean Urinary Free Cortisol (UFC) ≤ Upper Limit of Normal (ULN)
Description: The 24h-UFC concentration results from three samples during screening were averaged to obtain baseline. After baseline, mean 24h UFC was determined at week 24. At Week 4, 8, 16 and 20, mean 24h UFC was determined from two 24 hour urine collections collected on two consecutive days occurring before the visit. At Week 12, 24 and 48, the mean 24h-UFC from three 24 hour urine collections, collected over the week before the visit, was determined. After Week 24, the mean 24h UFC was determined at 12-week intervals until end of study visit, from two 24 hour collections during two consecutive days prior to each respective visit (except at Week 48). UFC was determined by liquid chromatography tandem mass spectroscopy (LC/MS/MS). The normal ranges were determined by the central laboratory's own reference range. All samples, including screening samples, were analyzed by a central laboratory.
Time Frame: Baseline, week 12, 24 and 48
Population: LOCF Week 24: last available mean 24h-UFC of at least two samples between and including week 12 and week 24; LOCF Week 48: last available mean 24h-UFC of at least two samples between and including week 12 and week 48. Two-sided 95% confidence intervals for proportions are calculated using the exact method
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pasireotide 600 μg: Pasireotide sub-cutaneous was supplied in 1 ml ampoules containing 600 μg pasireotide per 1 ml of solution and was administered BID. Starting dose was 600 μg for glucose impaired metabolism patients. Mean daily dose category is defined: 600 μg bid group includes all patients whose mean daily dose < 1500 μg /day.
- Pasireotide 900 μg: Pasireotide sub-cutaneous was supplied in 1 ml ampoules containing 900 μg pasireotide per 1 ml of solution and was administered BID. Starting dose was 900 μg. Mean daily dose category is defined : 900 μg bid group includes all patients whose mean daily dose ≥ 1500 μg /day
- All Patients: Patients received pasireotide 600 μg or 900 μg BID
Arm/Group | Pasireotide 600 μg | Pasireotide 900 μg | All Patients
Number analyzed (Participants) | 49 | 55 | 104
percentage of participants
  Week 12: number analyzed (Participants) | 27 | 39 | 66
  Week 12 | 77.8 [57.74 to 91.38] | 38.5 [23.36 to 55.38] | 54.5 [41.81 to 66.86]
  Week 24: number analyzed (Participants) | 22 | 24 | 46
  Week 24 | 68.2 [45.13 to 86.14] | 29.2 [12.62 to 51.09] | 47.8 [32.89 to 63.05]
  Week 48: number analyzed (Participants) | 10 | 11 | 21
  Week 48 | 70.0 [34.75 to 93.33] | 18.2 [2.28 to 51.78] | 42.9 [21.82 to 65.98]
  Week 24 (LOCF): number analyzed (Participants) | 37 | 49 | 86
  Week 24 (LOCF) | 54.1 [36.92 to 70.51] | 28.6 [16.59 to 43.26] | 39.5 [29.15 to 50.66]
  Week 48 (LOCF): number analyzed (Participants) | 37 | 49 | 86
  Week 48 (LOCF) | 51.4 [34.40 to 68.08] | 22.4 [11.78 to 36.62] | 34.9 [24.92 to 45.92]

3. Secondary Outcome: Percentage of Patients Achieving a Reduction of Mean UFC ≥ 50% From Baseline
Description: as for outcome 2
Time Frame: Baseline, week 12, 24 and 48
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pasireotide 600 μg | Pasireotide 900 μg | All Patients
Number analyzed (Participants) | 49 | 55 | 104
percentage of participants
  Week 12: number analyzed (Participants) | 27 | 39 | 66
  Week 12 | 74.1 [53.72 to 88.89] | 48.7 [32.42 to 65.22] | 59.1 [46.29 to 71.05]
  Week 24: number analyzed (Participants) | 22 | 24 | 46
  Week 24 | 68.2 [45.13 to 86.14] | 33.3 [15.63 to 55.32] | 50.00 [34.90 to 65.10]
  Week 48: number analyzed (Participants) | 10 | 11 | 21
  Week 48 | 60.0 [26.24 to 87.84] | 54.5 [23.38 to 83.25] | 57.1 [34.02 to 78.18]
  Week 24 (LOCF): number analyzed (Participants) | 37 | 49 | 86
  Week 24 (LOCF) | 56.8 [39.49 to 72.90] | 38.8 [25.20 to 53.76] | 46.5 [35.68 to 57.59]
  Week 48 (LOCF): number analyzed (Participants) | 37 | 49 | 86
  Week 48 (LOCF) | 51.4 [34.40 to 68.08] | 42.9 [28.82 to 57.79] | 46.5 [35.68 to 57.59]

4. Secondary Outcome: Percent Change in Cushing Quality of Life and Work Productivity and Activity Impairment-General Health (WPAI-GH) Scores
Description: A 12-item Cushing's syndrome HRQoL questionnaire (CushingQoL, cf. Webb et al 2008) was implemented and patients who completed 9 or more items at a visit were considered evaluable for that visit. The standardized scores were calculated as follows: 1) Obtain raw scores, denoted by X, as the sum of all the ratings on all the HRQoL questions for a single patient and the score can range from 12 (worst HRQoL) to 60 points (best HRQoL). Therefore, the lower the score, greater the negative impact on HRQoL and 2) obtain standardized score, Y, for a single patient
  • Y = 100 (X-12) / (60-12) = 100 (X-12)/48. For example, if a patient answers all 12 items with 'Sometimes' or 'Somewhat', X = 36 and Y = 100 ∙ 24/48 = 50 The WPAI-GH questionnaire was used to assess work productivity and activity impairment. However, there was very limited baseline data and therefore the results and outcomes of the objective, 'change from baseline in WPAI-GH scores' are not included.
Time Frame: Baseline, week 12, 24 and 48
Population: Only patients who completed at least 9 questions on questionnaire were included for that visit.
Measure: Mean (Standard Deviation); unit: percent change in score
Arm/Group | Pasireotide 600 μg | Pasireotide 900 μg | All Patients
Number analyzed (Participants) | 47 | 54 | 101
percent change in score
  Week 12: number analyzed (Participants) | 33 | 45 | 78
  Week 12 | 21.3 (47.03) | 100.8 (252.25) | 67.1 (197.09)
  Week 24: number analyzed (Participants) | 23 | 28 | 51
  Week 24 | 36.7 (59.25) | 119.7 (321.61) | 82.3 (243.19)
  Week 48: number analyzed (Participants) | 15 | 20 | 35
  Week 48 | 24.0 (37.76) | 42.3 (60.75) | 34.4 (52.29)

5. Secondary Outcome: Percent Change in Cushing's Disease Clinical Signs and Symptoms - Blood Pressure (BP)
Description: Standing systolic and diastolic BP based on 1 assessment and sitting systolic and diastolic BP was mean of 3 assessments.
Time Frame: Baseline, week 12, 24 and 48
Population: Number of patients with available data differed at visits
Measure: Mean (Standard Deviation); unit: percent change of mmhg
Arm/Group | Pasireotide 600 μg | Pasireotide 900 μg | All Patients
Number analyzed (Participants) | 49 | 55 | 104
percent change of mmhg
  Sitting systolic Week 12: number analyzed (Participants) | 35 | 45 | 80
  Sitting systolic Week 12 | -6.8 (12.04) | -1.4 (14.40) | -3.8 (13.61)
  Sitting systolic Week 24: number analyzed (Participants) | 24 | 29 | 53
  Sitting systolic Week 24 | -7.4 (8.97) | -5.7 (11.09) | -6.5 (10.13)
  Sitting systolic Week 48: number analyzed (Participants) | 16 | 21 | 37
  Sitting systolic Week 48 | -5.1 (8.57) | -4.7 (12.55) | -4.9 (10.87)
  Standing systolic Week 12: number analyzed (Participants) | 34 | 44 | 78
  Standing systolic Week 12 | -7.9 (12.49) | -3.6 (15.38) | -5.5 (14.27)
  Standing systolic Week 24: number analyzed (Participants) | 23 | 29 | 52
  Standing systolic Week 24 | -10.9 (10.30) | -6.7 (14.09) | -8.6 (12.62)
  Standing systolic Week 48: number analyzed (Participants) | 15 | 21 | 36
  Standing systolic Week 48 | -6.5 (9.45) | -4.4 (13.86) | -5.3 (12.10)
  Sitting diastolic Week 12: number analyzed (Participants) | 35 | 45 | 80
  Sitting diastolic Week 12 | -4.6 (15.13) | -0.2 (14.40) | -2.1 (14.79)
  Sitting diastolic Week 24: number analyzed (Participants) | 24 | 29 | 53
  Sitting diastolic Week 24 | -6.2 (7.29) | -3.8 (15.83) | -4.9 (12.65)
  Sitting diastolic Week 48: number analyzed (Participants) | 16 | 21 | 37
  Sitting diastolic Week 48 | -3.3 (10.38) | -4.3 (13.93) | -3.8 (12.37)
  Standing diastolic Week 12: number analyzed (Participants) | 34 | 44 | 78
  Standing diastolic Week 12 | -5.5 (16.02) | -1.9 (17.63) | -3.5 (16.93)
  Standing diastolic Week 24: number analyzed (Participants) | 23 | 29 | 52
  Standing diastolic Week 24 | -7.6 (10.30) | -5.3 (16.74) | -6.3 (14.18)
  Standing diastolic Week 48: number analyzed (Participants) | 15 | 21 | 36
  Standing diastolic Week 48 | -2.1 (13.78) | -4.4 (14.13) | -3.4 (13.83)

6. Secondary Outcome: Percent Change in Cushing's Disease Clinical Signs and Symptoms - Pulse
Description: Change from baseline is shown as: Percent change from baseline (BL) =((Post BL value - BL value)/ BL value)*100
Time Frame: Baseline, week 12, 24 and 48
Population: Number of patients with available data differed at visits
Measure: Mean (Standard Deviation); unit: percent change in bpm
Arm/Group | Pasireotide 600 μg | Pasireotide 900 μg | All Patients
Number analyzed (Participants) | 49 | 55 | 104
percent change in bpm
  Sitting pulse Week 12: number analyzed (Participants) | 35 | 45 | 80
  Sitting pulse Week 12 | 2.3 (18.93) | -7.5 (11.50) | -3.2 (15.87)
  Sitting pulse Week 24: number analyzed (Participants) | 24 | 29 | 53
  Sitting pulse Week 24 | -1.8 (17.05) | -2.6 (18.07) | -2.2 (17.46)
  Sitting pulse Week 48: number analyzed (Participants) | 16 | 21 | 37
  Sitting pulse Week 48 | 2.9 (16.39) | 3.7 (15.46) | 3.3 (15.65)

7. Secondary Outcome: Percent Change in Cushing's Disease Clinical Signs and Symptoms - Temperature
Description: degrees celius
Time Frame: Baseline week 12, 24 and 48
Population: Number of patients with available data differed at visits
Measure: Mean (Standard Deviation); unit: percent change in celius
Arm/Group | 600 µg Bid - All Grades | 900 μg - All Grades | All Patients - All Grades
Number analyzed (Participants) | 49 | 55 | 104
percent change in celius
  Week 12: number analyzed (Participants) | 33 | 43 | 76
  Week 12 | 0.1 (1.26) | -0.3 (1.06) | -0.1 (1.17)
  Week 24: number analyzed (Participants) | 21 | 28 | 49
  Week 24 | -0.1 (1.15) | -0.1 (1.26) | -0.1 (1.20)
  Week 48: number analyzed (Participants) | 15 | 20 | 35
  Week 48 | 0.03 (1.47) | -0.1 (1.19) | 0.1 (1.31)

8. Secondary Outcome: Percent Change in Cushing's Disease Clinical Signs and Symptoms - Body Mass Index (BMI)
Description: Percent change in patients reducing by at least one class level. Class levels: <25.0, 25.0 to <30.0, ≥ 30.0. Percent change from baseline (BL) =((Post BL value - BL value)/ BL value)*100
Time Frame: Baseline, week 12, 24 and 48
Population: Number of patients with available data differed at visits
Measure: Mean (Standard Deviation); unit: percent change in kg/m2
Arm/Group | Pasireotide 600 μg | Pasireotide 900 μg | All Patients
Number analyzed (Participants) | 49 | 55 | 104
percent change in kg/m2
  Week 12: number analyzed (Participants) | 35 | 44 | 79
  Week 12 | -4.2 (3.70) | -4.8 (5.38) | -4.5 (4.69)
  Week 24: number analyzed (Participants) | 24 | 29 | 53
  Week 24 | -7.3 (5.46) | -5.2 (6.51) | -6.1 (6.10)
  Week 48: number analyzed (Participants) | 16 | 21 | 37
  Week 48 | -8.0 (6.82) | -6.3 (7.88) | -7.0 (7.39)

9. Secondary Outcome: Percent Change in Cushing's Disease Clinical Signs and Symptoms - Weight
Description: Clinically relevant threshold (at any time point) was reduction of ≥ 5%
Time Frame: Baseline, week 12, 24 and 48
Population: Number of patients with available data differed at visits
Measure: Mean (Standard Deviation); unit: percent change in kg
Arm/Group | Pasireotide 600 μg | Pasireotide 900 μg | All Patients
Number analyzed (Participants) | 49 | 55 | 104
percent change in kg
  Week 12: number analyzed (Participants) | 35 | 44 | 79
  Week 12 | -4.2 (3.70) | -4.8 (5.38) | -4.5 (4.69)
  Week 24: number analyzed (Participants) | 24 | 29 | 53
  Week 24 | -7.3 (5.46) | -5.2 (6.51) | -6.1 (6.10)
  Week 48: number analyzed (Participants) | 16 | 21 | 37
  Week 48 | -8.0 (6.82) | -6.3 (7.88) | -7.0 (7.39)

10. Secondary Outcome: Percent Change in Cushing's Disease Clinical Signs and Symptoms - Muscle Strength
Description: Direct observation of ability to stand unaided: 0=able to stand easily with arms extended, 1=able to stand after several efforts without using arms as assistance, 2=able to stand only by using arms as assistance 3=completely unable to stand
Time Frame: Baseline, week 12, 24 and 48
Population: Number of patients with available data differed at visits
Measure: Mean (Standard Deviation); unit: percent change in scores
Arm/Group | Pasireotide 600 μg | Pasireotide 900 μg | All Patients
Number analyzed (Participants) | 49 | 55 | 104
percent change in scores
  Week 12: number analyzed (Participants) | 13 | 9 | 22
  Week 12 | -34.6 (62.53) | -53.7 (46.98) | -42.4 (56.28)
  Week 24: number analyzed (Participants) | 7 | 7 | 14
  Week 24 | -28.6 (48.80) | -47.6 (50.40) | -38.1 (48.67)
  Week 48: number analyzed (Participants) | 5 | 4 | 9
  Week 48 | -30.0 (44.72) | -75.0 (50.0) | -50.0 (50.00)

11. Secondary Outcome: Percent Change in Cushing's Disease Clinical Signs and Symptoms - Waist Circumference
Description: Clinically relevant threshold (at any time point). Reduction of ≥ 5%, Reduction of ≥ 10%
Time Frame: Baseline, week 12, 24 and 48
Population: Number of patients with available data differed at visits
Measure: Mean (Standard Deviation); unit: percent change of centimeters
Arm/Group | Pasireotide 600 μg | Pasireotide 900 μg | All Patients
Number analyzed (Participants) | 49 | 55 | 104
percent change of centimeters
  Week 12: number analyzed (Participants) | 35 | 42 | 77
  Week 12 | -2.0 (4.29) | -2.9 (6.70) | -2.5 (5.72)
  Week 24: number analyzed (Participants) | 24 | 28 | 52
  Week 24 | -5.8 (6.28) | -3.1 (5.48) | -4.4 (5.96)
  Week 48: number analyzed (Participants) | 16 | 20 | 36
  Week 48 | -5.1 (5.74) | -4.1 (5.64) | -4.6 (5.62)

12. Secondary Outcome: Percent Change in Cushing's Disease Clinical Signs and Symptoms - Hirsutism
Description: Change from baseline is shown as: Percent change from baseline (BL) =((Post BL value - BL value)/ BL value)*100. Ferriman-Gallway scoring was used: 0=minimum and 36 was maximum in females only.
Time Frame: Baseline, week 12, 24 and 48
Population: Number of patients with available data differed at visits
Measure: Mean (Standard Deviation); unit: percent change in scores
Arm/Group | Pasireotide 600 μg | Pasireotide 900 μg | All Patients
Number analyzed (Participants) | 37 | 47 | 84
percent change in scores
  Week 12: number analyzed (Participants) | 24 | 31 | 55
  Week 12 | -12.2 (24.57) | -8.2 (35.30) | -10.0 (30.88)
  Week 24: number analyzed (Participants) | 16 | 20 | 36
  Week 24 | -21.2 (32.72) | -16.2 (46.99) | 18.4 (40.79)
  Week 48: number analyzed (Participants) | 11 | 15 | 26
  Week 48 | -18.2 (30.12) | 9.6 (143.83) | -2.2 (110.20)

13. Secondary Outcome: Percent Change From Baseline in Growth Hormone (GH) Values
Description: Descriptive summary of the effect of pasireotide on GH.
Time Frame: Baseline, week 12, 24 and 48
Population: Number of patients with available data differed at visits
Measure: Mean (Standard Deviation); unit: percent change of µg/L
Arm/Group | Pasireotide 600 μg | Pasireotide 900 μg | All Patients
Number analyzed (Participants) | 48 | 55 | 103
percent change of µg/L
  Week 12: number analyzed (Participants) | 35 | 45 | 80
  Week 12 | -17.3 (109.89) | -20.90 (156.60) | -19.3 (137.33)
  Week 24: number analyzed (Participants) | 22 | 29 | 51
  Week 24 | -22.2 (62.43) | -26.2 (105.44) | -24.4 (88.70)
  Week 48: number analyzed (Participants) | 16 | 20 | 36
  Week 48 | 23.1 (127.30) | -1.0 (134.97) | 9.7 (130.32)

14. Secondary Outcome: Percent Change From Baseline in Insulin Growth Factor - 1 (IGF - 1) Values
Description: Descriptive summary of the effect of pasireotide on IGF-1
Time Frame: Baseline, week 12, 24 and 48
Population: Number of patients with available data differed at visits
Measure: Mean (Standard Deviation); unit: percent change of ng/ml
Arm/Group | Pasireotide 600 μg | Pasireotide 900 μg | All Patients
Number analyzed (Participants) | 48 | 53 | 101
percent change of ng/ml
  Week 12: number analyzed (Participants) | 34 | 44 | 78
  Week 12 | -53.4 (23.66) | -57.8 (23.93) | -55.9 (23.76)
  Week 24: number analyzed (Participants) | 23 | 29 | 52
  Week 24 | -49.2 (26.56) | -56.2 (26.55) | -53.1 (26.53)
  Week 48: number analyzed (Participants) | 16 | 21 | 37
  Week 48 | -41.8 (35.72) | -52.1 (21.87) | -47.6 (28.71)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit up to approximately 256 weeks
Description: Consistent with EudraCT disclosure specifications, Novartis has reported under the Serious adverse events fields "number of deaths resulting from adverse events" all those deaths, resulting from serious adverse events that are deemed to be causally related to treatment by the investigator
Groups:
- 600 µg Bid: 600 µg bid
- 900 µg Bid: 900 µg bid
- All Patients: All patients
Arm/Group | 600 µg Bid | 900 µg Bid | All Patients
All-Cause Mortality (participants affected / at risk) | 0/49 | 1/55 | 1/104
Serious Adverse Events (participants affected / at risk) | 13/49 | 17/55 | 30/104
Other Adverse Events (participants affected / at risk) | 49/49 | 54/55 | 103/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 600 µg Bid (N=49) | 900 µg Bid (N=55) | All Patients (N=104)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 1
Glucocorticoid deficiency (Endocrine disorders) | 1 | 0 | 1
Hyperprolactinaemia (Endocrine disorders) | 1 | 0 | 1
Pituitary-dependent Cushing's syndrome (Endocrine disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 3
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 0 | 1
Death (General disorders) | 0 | 1 | 1
Drug ineffective (General disorders) | 0 | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 3 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic lesion (Hepatobiliary disorders) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1
Dengue fever (Infections and infestations) | 1 | 0 | 1
Meningitis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Blood cortisol increased (Investigations) | 1 | 0 | 1
Lipase abnormal (Investigations) | 1 | 0 | 1
Transaminases increased (Investigations) | 1 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Embolism venous (Vascular disorders) | 0 | 1 | 1
Venous thrombosis (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 600 µg Bid (N=49) | 900 µg Bid (N=55) | All Patients (N=104)
Bradycardia (Cardiac disorders) | 2 | 3 | 5
Sinus bradycardia (Cardiac disorders) | 4 | 1 | 5
Adrenal insufficiency (Endocrine disorders) | 4 | 1 | 5
Hypothyroidism (Endocrine disorders) | 3 | 1 | 4
Abdominal discomfort (Gastrointestinal disorders) | 1 | 3 | 4
Abdominal pain (Gastrointestinal disorders) | 10 | 9 | 19
Abdominal pain upper (Gastrointestinal disorders) | 2 | 6 | 8
Constipation (Gastrointestinal disorders) | 1 | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 28 | 23 | 51
Dry mouth (Gastrointestinal disorders) | 5 | 3 | 8
Dyspepsia (Gastrointestinal disorders) | 2 | 4 | 6
Faeces soft (Gastrointestinal disorders) | 4 | 1 | 5
Flatulence (Gastrointestinal disorders) | 6 | 5 | 11
Frequent bowel movements (Gastrointestinal disorders) | 3 | 2 | 5
Nausea (Gastrointestinal disorders) | 22 | 26 | 48
Vomiting (Gastrointestinal disorders) | 3 | 7 | 10
Asthenia (General disorders) | 4 | 7 | 11
Fatigue (General disorders) | 11 | 12 | 23
Injection site erythema (General disorders) | 3 | 2 | 5
Oedema peripheral (General disorders) | 9 | 3 | 12
Cholelithiasis (Hepatobiliary disorders) | 8 | 22 | 30
Hepatic steatosis (Hepatobiliary disorders) | 1 | 4 | 5
Gastroenteritis (Infections and infestations) | 3 | 2 | 5
Influenza (Infections and infestations) | 1 | 3 | 4
Nasopharyngitis (Infections and infestations) | 2 | 7 | 9
Upper respiratory tract infection (Infections and infestations) | 1 | 6 | 7
Urinary tract infection (Infections and infestations) | 0 | 4 | 4
Procedural nausea (Injury, poisoning and procedural complications) | 3 | 5 | 8
Procedural pain (Injury, poisoning and procedural complications) | 0 | 3 | 3
Alanine aminotransferase increased (Investigations) | 3 | 1 | 4
Blood cortisol decreased (Investigations) | 3 | 1 | 4
Blood glucose increased (Investigations) | 4 | 9 | 13
Electrocardiogram QT prolonged (Investigations) | 3 | 1 | 4
Gamma-glutamyltransferase increased (Investigations) | 3 | 4 | 7
Insulin-like growth factor decreased (Investigations) | 5 | 5 | 10
Weight decreased (Investigations) | 3 | 2 | 5
Decreased appetite (Metabolism and nutrition disorders) | 6 | 1 | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 9 | 14 | 23
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 3 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 19 | 22 | 41
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 3 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 4
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 5 | 3 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 3 | 8
Dizziness (Nervous system disorders) | 6 | 8 | 14
Headache (Nervous system disorders) | 12 | 19 | 31
Presyncope (Nervous system disorders) | 3 | 1 | 4
Syncope (Nervous system disorders) | 3 | 0 | 3
Anxiety (Psychiatric disorders) | 2 | 3 | 5
Depression (Psychiatric disorders) | 4 | 3 | 7
Insomnia (Psychiatric disorders) | 1 | 4 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 7 | 11
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 4 | 6
Hypertension (Vascular disorders) | 3 | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/61/NCT01582061/SAP_000.pdf
  • Study Protocol (2015-11-13): https://cdn.clinicaltrials.gov/large-docs/61/NCT01582061/Prot_001.pdf